CLINICAL TRIAL: NCT05821686
Title: Efficacy of Intralesional IL-2 for Resectable Triple Negative Breast Cancer
Brief Title: Efficacy of Interleukin-2 in Triple Negative Breast Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IL-2.001
Record Dates: First submitted 2022-11-18; First posted 2023-04-20 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-08

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Intralesional IL-2 therapy x 4 weeks between initial consultation and planned surgery
  Interventions: Drug: Human Interleukin-2 (IL-2) (Proleukin)

INTERVENTIONS:
Drug: Human Interleukin-2 (IL-2) (Proleukin) — All the recruited participants will receive 4 intralesional injections of Interleukin-2 with a dose of 500,000 international units (IU) per mm width of tumor to max dose of 10 million IU.

SUMMARY:
This study is a single arm, phase II pilot design. The study will evaluate the safety and efficacy of intralesional immunotherapy (e.g. IL-2) in early stage TNBC. The overall objective of the research study is to advance our knowledge of novel immunotherapies and routes of administration for the treatment of TNBC

HYPOTHESES: Neoadjuvant treatment of TNBC with intralesional IL-2 is safe and well tolerated and can produce a pathological response.

Aim 1: Examine the safety and possible efficacy of a novel neoadjuvant intralesional intervention (IL-2) for patients with early-stage TNBC.

DETAILED DESCRIPTION:
Breast cancer is a leading cause of cancer related death in women. Triple negative breast cancer (TNBC) is a subtype of breast cancer based on an immunohistochemistry that lacks estrogen receptor (ER), progesterone receptor (PR) and human epidermal growth factor-2 (HER2) expression. It is known to disproportionately affects younger women and women of African ancestry. TNBCs account for approximately 15-20% of all newly diagnosed breast cancer. Compared to other subtypes of breast cancer, including hormone sensitive disease, TNBC is associated with a high risk of distant metastases and is associated with a lower disease-free and overall survival. As TNBCs lack expression for ER, PR and HER-2, targeted therapies are ineffective. Immunotherapy has emerged as an important treatment strategy in TNBC. Traditionally, breast cancer has been considered a 'cold' cancer but the disease is highly heterogenous and TNBC appears to be more immunogenic (i.e. 'hot'). Compared to other forms of the disease, TNBC is associated with a higher mutational burden, tumor infiltrating lymphocytes (TILs) and PD-L1 expression. The later is associated with response to immunotherapy. Indeed, systemic immunotherapy is now approved as first line therapy for metastatic and unresectable PD-L1 positive TNBC. Systemic immunotherapy may also increase the incidence of pathologic complete response after neoadjuvant therapy in early stage TNBC. Improvement in pathologic complete response is weighed against rare but life-threatening immune related side-effects of immunotherapy, including adrenal insufficiency, pneumonitis causing respiratory arrest and multi-organ dysfunction syndrome.

Interleukin-2 is one of the first immunomodulating agents to be approved for cancer treatment, including renal cell carcinoma and melanoma. The cytokine plays an important role in the maintenance CD4+ regulatory T-cells and the differentiation of CD4+ T-cells into a variety of subsets. It also promotes CD8+ T-cell and NK cell cytotoxicity activity and modulates T-cell differentiation in response to antigen presentation. Systemically, IL-2 is limited by a short half-life and significant toxicities. The intralesional injection of IL-2 eliminates the undesirable grade II/III toxicities and often severe side effects of the therapy, while achieving high doses of IL-2 at the tumor site. The most common side effect of intralesional IL-2 is inflammation at the site of injection and mild flu like symptoms, including fatigue and nausea. Rarely patients may experience low-grade fever or headache, which are easily controlled by over-the-counter medications. A number of studies have reported on the use of intralesional IL-2 in management of in-transit melanoma. In this patient population, intralesional IL-2 produces a durable complete response. Much less has been published on its use in other cancers, such as breast cancer. However, there is case report level evidence to suggest that intralesional IL-2 can produce a pathologic complete response in metastatic / unresectable TNBC.

The present study considers the significant scope that remains to improve the outcomes for women with TNBC. This study seeks to build upon the growing body of evidence in support of immunomodulation in the treatment of TNBC, while also exploring a different and less toxic route of administration (i.e. intralesional as opposed to systemic). In the window of opportunity between the time of initial surgical consultation and planned OR for patients proceeding with upfront surgery, this study proposes to provide intralesional IL-2 with immediate pathologic assessment.

This 'window of opportunity' design will provide us opportunity to conduct a pilot study to evaluate the efficacy of an intralesional immunotherapy (e.g. IL-2) in early stage TNBC as a well-tolerated, low-risk intervention with the potential to improve outcomes without the toxicity of systemic treatment. As systemic immunotherapy moves from the metastatic setting to the adjuvant setting and is increasingly being used in earlier and earlier stage disease, the rationale for systemic therapy with systemic side effects to treat a local disease becomes harder to justify. This study seeks to challenge the notion that the only effective immunotherapy in the treatment of TNBC is systemic and perhaps a local administration can produce the immune response needed to affect significant pathologic response.

ELIGIBILITY:
Inclusion Criteria:

1. Women with biopsy proven TNBC who are not scheduled to receive neoadjuvant chemotherapy.
2. Tumors ≤ 2 cm (clinical T1N0)
3. Planned upfront surgery (patient preference)
4. Medically unable to receive neoadjuvant chemotherapy
5. 18 - 80 years of age.
6. Able to provide consent for the study.
7. Able to come to the hospital for the intralesional injections.

Exclusion Criteria:

1. No diagnosis of TNBC.
2. Not able to provide consent for the study.
3. Not able to come to the hospital for study visits.
4. Presence of any contraindication for IL-2 therapy (abnormal thallium stress test, abnormal pulmonary function test, organ allograft and toxicities with a previous dosage).
5. Participant has experienced IL-2 related toxicities during an earlier course of therapy (sustained ventricular tachycardia; cardiac arrythmias unresponsive to management; chest pain with ECG changes consistent with angina or myocardial infarction; cardiac tamponade; intubation required > 72 hours; renal failure requiring dialysis > 72 hours; coma, or toxic psychosis > 48 hours; repetitive or difficult to control seizures; bowel ischemia; gastrointestinal bleeding requiring surgery)
6. If participant is on cancer treatment drugs and steroids to avoid drug interactions.
7. Known pregnancy and breast feeding. There are no known studies to support the use of interleukin in pregnancy and breast-feeding mothers.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Pathologic response as defined by the residual cancer burden (RCB) index (RCB 0-IV) | measured immediately after surgery during routine pathological assessment
  Presence of in-situ disease alone will be considered a pCR

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of intralesional IL-2 | 1 year
  The number of patients experiencing an adverse event will be defined and quantified (i.e. severity) using the Common Terminology Criteria for Adverse Events during treatment with intralesional IL-2
Proportion of Patients who Complete 4 cycles of Intralesional IL-2 | 1 year
  What percentage of patients who are enrolled complete all 4 intended cycles if intralesional IL-2. Only patients who are enrolled and receive at least 1 cycle will be included in the denominator.

IPD SHARING:
Plan to Share IPD: No